CLINICAL TRIAL: NCT03765294
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Study to Investigate the Effects of ACT-541468 on Nighttime Respiratory Function in Patients With Mild to Moderate Obstructive Sleep Apnea
Brief Title: A Study to Investigate the Effects of ACT-541468 on Nighttime Respiratory Function in Patients With Mild to Moderate Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078-110; 2018-002360-96 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: 2-way cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: ACT-541468 (Experimental): 50 mg once daily from Day 1 to Day 5 of Period A
  Interventions: Drug: ACT-541468
- Treatment B: Placebo (Placebo Comparator): Matching placebo once daily from Day 1 to Day 5 of Period B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-541468 — Film-coated tablet for oral use
  Arms: Treatment A: ACT-541468
Drug: Placebo — Film-coated tablet for oral use
  Arms: Treatment B: Placebo

SUMMARY:
This study is conducted to investigate the effects of ACT-541468 on nighttime respiratory function in patients with mild to moderate obstructive sleep apnea

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Male and female subjects aged ≥ 18 years at Screening.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Screening Visit 2 and on Day 1 pre-dose of the first period. They must agree to consistently and correctly use a highly effective method of contraception with a failure rate of < 1% per year.
* Women of non-childbearing potential, i.e., postmenopausal, with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure, XY genotype, Turner syndrome, and/or uterine agenesis.
* Diagnosis of OSA according to the International Classification of Sleep Disorders documented by medical history and confirmed in a sleep laboratory in the context of diagnosing OSA within the last 3 years.
* Patient with mild to moderate intensity of OSA determined during OSA diagnosis and confirmed on the screening night PSG and defined as apnea/hypopnea index (AHI) ranging from 5 to < 30.

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Pregnant or lactating women.
* Modified Swiss Narcolepsy Scale total score < 0 at Screening, or history of narcolepsy or cataplexy.
* Subjects with clinically significant abnormality on the screening night PSG as per investigator judgment, including evidence of severe insomnia (i.e., sleep time < 5 h) periodic limb movement disorder with arousal index ≥ 10/h, restless legs syndrome, circadian rhythm disorder, REM behavior disorder, parasomnia including nightmare disorder, sleep terror disorder, and/or sleepwalking disorder.
* Need for continuous positive airway pressure device or a dental appliance device within the preceding 7 days prior to Screening Visit 2 and during the course of the study, i.e., from Screening Visit 2 to EOS.
* Evidence of any other clinically significant active pulmonary disease such as chronic obstructive pulmonary disease (COPD) (as per Global Initiative for Obstructive Lung Disease), based on investigator's judgment.
* History of surgical intervention for obstructive sleep apnea, except nose surgery.
* SaO2 < 90% during wakefulness or mean non-apneic SaO2 (i.e., outside events of apnea/hypopnea) < 85% for > 5 consecutive min during the screening night PSG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Apnea/hypopnea index (AHI) after multiple-dose administration of ACT-541468 as measured by polysomnography (PSG) | After multiple-dose administration (i.e., at Night 5) (duration: 8 hours PSG recording)
  AHI is defined by total number of apnea (pause in respiration ≥ 10 s) plus hypopnea (reduction in airflow or tidal volume from pre-event baseline by 30% for at least 10 s accompanied by a decrease of SaO2 ≥ 4%) events, divided by total sleep time (TST, in min), then multiplied by 60, during TST

OTHER OUTCOMES:
AHI during TST after single-dose administration | After single-dose (i.e., Night 1) administration (duration: 8 hours PSG recording)
Mean SaO2 during TST | After single-dose (i.e., Night 1) administration (duration: 8 hours PSG recording)
AHI during the awake, non-REM, and REM phases | After single-dose (i.e., Night 1) administration (duration: 8 hours PSG recording)
Mean SaO2 during the awake, non-REM, and REM phases | After single-dose (i.e., Night 1) administration (duration: 8 hours PSG recording)
Percentage of TST during which SaO2 is < 90%, < 85%, and < 80% | After single-dose (i.e., Night 1) administration (duration: 8 hours PSG recording)
Change from baseline to EOP of both periods in subjective next-day performance (morning sleepiness, daytime alertness, and daytime ability to function) as assessed by VAS | After single-dose (i.e., Night 1) and multiple-dose (i.e., Night 5) administration (duration: 2 x 8 hours PSG recording)
Objective sleep parameters LPS, WASO, TST, and SEI following single- and multiple-dose administration, as measured by PSG | After single-dose (i.e., Night 1) and multiple-dose (i.e., Night 5) administration (duration: 2 x 8 hours PSG recording)
Safety profile including incidence of adverse events (AEs) and serious adverse events (SAEs) | From baseline to EOS (duration: for up to 10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Advanced Sleep Research, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boof ML, Ufer M, Fietze I, Pepin JL, Guern AS, Lemoine V, Dingemanse J. Assessment of the effect of the dual orexin receptor antagonist daridorexant on various indices of disease severity in patients with mild to moderate obstructive sleep apnea. Sleep Med. 2022 Apr;92:4-11. doi: 10.1016/j.sleep.2021.11.015. Epub 2022 Feb 12. PMID 35306405
- [Derived] Boof ML, Dingemanse J, Lederer K, Fietze I, Ufer M. Effect of the new dual orexin receptor antagonist daridorexant on nighttime respiratory function and sleep in patients with mild and moderate obstructive sleep apnea. Sleep. 2021 Jun 11;44(6):zsaa275. doi: 10.1093/sleep/zsaa275. PMID 33305817